CLINICAL TRIAL: NCT04771052
Title: Minimizing the Effects of COVID-19 Hospitalization With the COVID Rehabilitation Program for the Elderly: the CORE Trial in Response to the Pandemic
Brief Title: Minimizing the Effects of COVID-19 Hospitalization With the COVID Rehabilitation Program for the Elderly
Acronym: CORE
Status: Completed | Type: Observational
Sponsor: Université de Sherbrooke (Other)
Responsible Party: Sponsor
Other Study IDs: MP-31-2021-3770
Record Dates: First submitted 2021-02-23; First posted 2021-02-25 (Actual); Last update posted 2022-05-23 (Actual); Status verified 2022-05

CONDITIONS: Covid19
MeSH Terms: conditions — COVID-19

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Retrospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- CORE program: Patients admitted to a dedicated COVID-19 units (CHUS Hôtel-Dieu de Sherbrooke - CIUSSS de L'Estrie - CHUS) with medical clearance (physical deconditioning; hemodynamically stable; oxygen therapy by nasal cannula < 4 L/min for saturation > 92%; resting respiratory rate < 24; and heart rate between 50 and 120 beats per minute).
  Interventions: Other: COVID Rehabilitation Program for the Elderly (CORE)
- Control: Patients admitted to a dedicated COVID-19 units (CHAUR de Trois-Rivières, CIUSSS de la Mauricie-et-du-Centre-du-Québec) receiving usual care, matched to CORE a patient with similar characteristics (sex, age, preadmission provenance).

INTERVENTIONS:
Other: COVID Rehabilitation Program for the Elderly (CORE) — In the intervention unit, two teams (core team: physiotherapists and service healthcare workers; specialized team: occupational therapist, registered dietician, social worker) are dedicated to the patients hospitalized in COVID-19 unit. To prevent malnutrition, caused by disease-associated inflammation, the Nutrition as Medicine program (prescribed small doses (30 or 60 mL; 2 kcal/mL) of oral nutrition supplement dispensed with medication pass, 1 to 4 times a day), has been systematically implemented (collective prescription). To improve muscle strength, balance and tissue oxygenation and concomitantly reduce immobilization and risk of falls, each patient has a private pedal exerciser, resistance elastic bands and free weights to perform a progressive, monitored and individualized rehabilitation program thrice a day.
  Groups: CORE program

SUMMARY:
Although evidence from the management of other viral respiratory infections suggest that early multidisciplinary rehabilitation could mitigate the adverse effects of the severe form of the illness, and reduce the length of hospital stays (LOS), specific data for COVID-19 are lacking. Hence, in response to the current pandemic, we propose to implement and assess the impact of an early standardized multidisciplinary rehabilitation program tailored to frail older adults on 1) LOS, 2) post-discharge destination, 3) prognostic index and 4) functional capacity.

With a pragmatic multicenter controlled study, the COvid Rehabilitation Program for the Elderly (CORE) trial will allow to measure the effectiveness of a multidisciplinary program to minimize the effects of hospitalization and provide the required tools to rapidly implement an innovative strategy of care for older adults. Indeed, based on the results of this study, and with the support of scientific and professional organizations, a standardized program tailored to older adults with COVID-19 will be disseminated in Canada for all medical units dedicated to the management of the disease. Because of its pragmatic approach, this study will provide a sustainable multidisciplinary intervention that can be quickly implemented in any Canadian (or abroad) COVID-19 medical unit. Finally, given that COVID-19 is the third coronavirus infection in the last 20 years, the expected results will provide guidelines, with decision tree algorithms, for implementation should another coronavirus or for that matter, any other such type of infection that surface in the future.

ELIGIBILITY:
Inclusion Criteria:

* Patients with medical clearance (physical deconditioning; hemodynamically stable; oxygen therapy by nasal cannula < 4 L/min for saturation > 92%; resting respiratory rate < 24; and heart rate between 50 and 120 beats per minute). Controls were paired with those of the CORE program according to age, sex and pre-admission origin

Exclusion Criteria:

* None

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Study Population: Patients admitted to the COVID unit at CHUS Hôtel-Dieu de Sherbrooke - CIUSSS de L'Estrie - CHUS (CORE program) or CHAUR de Trois-Rivières, CIUSSS de la Mauricie-et-du-Centre-du-Québec (Controls)
Sampling Method: Non-Probability Sample
Enrollment: 124 (Actual)
Dates: Start 2020-09-01 (Actual); Primary Completion 2021-08-31 (Actual); Study Completion 2022-01-05 (Actual)

PRIMARY OUTCOMES:
Length of stay | 1 day after discharge
  Length of stay in COVID and subacute unit (days)

SECONDARY OUTCOMES:
Post-discharge destination | 1 day after discharge
  (home; long-term care facilities; death) or transfer to a specialized subacute unit (e.g., rehabilitation geriatric unit)
Readmission rate 30 days after discharge | 30 days after discharge
Change in patient prognosis | At baseline (± 2 days after admission in the COVID-19 unit) and before discharge (± 3 days)
  Evaluated using the COVID-19 vulnerability index (symptoms, medical history, and sociodemographic data)
Change in functional capacity (lower limb function) | At baseline (± 2 days after admission in the COVID-19 unit) and before discharge (± 3 days)
  Lower limb function is assessed using the 5-repetition sit-to-stand test (reported in seconds)
Change in functional capacity (handgrip strength) | At baseline (± 2 days after admission in the COVID-19 unit) and before discharge (± 3 days)
  Handgrip strength is measured using a handgrip dynamometer (reported in kg)

CONTACTS AND LOCATIONS:
Locations (2):
- Canada (2):
  - CIUSSS de l'Estrie-Centre hospitalier universitaire de Sherbrooke (CHUS), Sherbrooke, Quebec
  - Centre hospitalier affilié universitaire régional (CHAUR), Trois-Rivières, Quebec

IPD SHARING:
Plan to Share IPD: No